CLINICAL TRIAL: NCT04742946
Title: Digital Physiotherapy Practice in Long Covid-19 Patients to Improve Functional Capacity and Quality of Life.
Brief Title: Digital Physiotherapy Practice in Long Covid-19 Patients
Acronym: TRCovidA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universidad de Granada (Other)
Collaborators: University of Malaga (Other)
Responsible Party: Principal Investigator, María José Estebanez Pérez, Principal Investigator. PhD, University of Malaga
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRCovidAndalucía
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Long COVID-19 Syndrome
Keywords: Digital Physiotherapy Practice (Telerehabilitation); Covid19 sequelae
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Telerehabilitation; Telemedicine

STUDY DESIGN:
Intervention Model Description: A quasi-experimental pre-post study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TR Group (Experimental): Personalized digital physiotherapy program 4 weeks. One session per day. Web and mobile application. Auto-Exercise
  Interventions: Other: Digital Physiotherapy Practice (Telerehabilitation)

INTERVENTIONS:
Other: Digital Physiotherapy Practice (Telerehabilitation) — Online Physiotherapy services
  Other Names: Telemedicine, ehealth

SUMMARY:
The COVID-19 can cause important sequels in the respiratory system by bilateral pneumonia and frequently presents loss of strength, dyspnea, polyneuropathies and multi-organic affectation. Long COVID-19 has been defined as the condition occurring in individuals with a history of probable or confirmed SARS-CoV-2 infection, with related symptoms lasting at least 2 months and not explainable by an alternative diagnosis. The practice of digital physiotherapy presents itself as a promising complementary treatment method to standard physiotherapy, playing a key role in the recovery of function in subjects who have passed the disease and who maintain some symptomatology over time. The aims of this research are to explore the effect of a digital physiotherapy intervention on functional recovery in patients diagnosed with Long COVID-19 and to identify the level of adherence to the treatment carried out. Physiotherapy interventions acquires a fundamental role in the recovery of the functions and the quality of life. As secondary objectives, the aim is to identify the satisfaction and perception of patients with the intervention and the presence of barriers to its implementation (throught a qualitative research), as well as to evaluate the cost-effectiveness from the perspective of the health system. A quasi-experimental pre-post study assessed initially and at the end of the 4-week intervention the functional capacity (1-min STS and SPPB) and the adherence (software). The hypothesis of this research is that the implementation of a TR program presents positive results. If hypothesis is confirmed, that would be an opportunity to define new policies and interventions to address this disease and its consequences.

DETAILED DESCRIPTION:
The authors hypothesised that the implementation of a digital physiotherapy intervention in Long COVID-19 participants is effective to improve the functional capacity and adherence and have positive results in patients satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Adult over 18 years old
* Diagnosis: Long COVID-19 syndrome
* Residing in the Andalusian Community during the research period
* To have a computer technology with an internet connection aat home (personal computer, laptop, tablet or smartphone)
* Ability and knowledge to access email or whatsapp

Exclusion Criteria:

-Cognitive ability not suitable for the use of technological tools

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Functional Capacity | Baseline (T0)
  sit-to-stand test in 1 minute
Functional Capacity | 4 weeks (T1)
  sit-to-stand test in 1 minute
Functional Capacity (SPBB) short performance physical battery test | Baseline (T0)
  (SPBB) short performance physical battery test
Functional Capacity (SPBB) short performance physical battery test | Baseline 4 weeks (T1)
  (SPBB) short performance physical battery test
The Short Form Health Survey SF-12 | Baseline (T0)
  Quality of Live. For each of the 8 dimensions, the items are coded, aggregated and transformed into a scale ranging from 0 (the worst health status for that dimension) to 0 (the worst health status for that dimension).
  a scale ranging from 0 (the worst health status for that dimension) to 100 (the best health status).
  100 (the best health status)
The Short Form Health Survey SF-12 Quality of Live | 4 weeks (T1)
  The SF-12 For each of the 8 dimensions, the items are coded, aggregated and transformed into a scale ranging from 0 (the worst health status for that dimension) to 0 (the worst health status for that dimension).
  a scale ranging from 0 (the worst health status for that dimension) to 100 (the best health status).
  100 (the best health status)
European Quality of Life-5 Dimensions EQ-5D | Baseline (T0)
  Quality of Live The responses to the five EQ-5D dimensions (i.e. an EQ-5D health state or profile) can be converted into a single number called an index value. The index value reflects how good or bad the health state is according to the preferences of the general population of a country/region. The collection of index values for all possible EQ-5D states is called a value set. Value sets are currently available for the EQ-5D-3L and EQ-5D-5L for different countries/regions. Several valuation techniques have been used to generate these value sets: time trade-off (TTO), visual analogue scale (VAS), and more recently, discrete choice experiments (DCE).
European Quality of Life-5 Dimensions EQ-5D | 4 weeks (T1)
  Quality of Live The responses to the five EQ-5D dimensions (i.e. an EQ-5D health state or profile) can be converted into a single number called an index value. The index value reflects how good or bad the health state is according to the preferences of the general population of a country/region. The collection of index values for all possible EQ-5D states is called a value set. Value sets are currently available for the EQ-5D-3L and EQ-5D-5L for different countries/regions. Several valuation techniques have been used to generate these value sets: time trade-off (TTO), visual analogue scale (VAS), and more recently, discrete choice experiments (DCE).

SECONDARY OUTCOMES:
Telemedicine Satisfaction Questionnaire (TSQ) | 4 weeks (T1)
  Telemedicine Satisfaction Questionnaire (TSQ). Perceived satisfaction comparing telemedicine to inperson in 26 Questions with likert scales
Cost-effectiveness of the telerehabilitation intervention | 4 weeks T1
  Direct Costs
Adherence to intervention | 4 weeks T1
  Automatic register by the digital physiotherapy software. Number of treatments and exercise acoording to PT prescription.
Satisfaction and Perception with intervention | 4 weeks T1
  Qualitative interview

CONTACTS AND LOCATIONS:
Overall Officials: José-Manuel Pastora-Bernal, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- Facultad Ciencias de la Salud, Málaga, Spain

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, Statistical Analysis plan and outcomes measures will be shared
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 8 weeks
Access Criteria: data will be shared upon request to the principal investigator

REFERENCES:
- [Result] Del Rio C, Malani PN. 2019 Novel Coronavirus-Important Information for Clinicians. JAMA. 2020 Mar 17;323(11):1039-1040. doi: 10.1001/jama.2020.1490. No abstract available. PMID 32022836
- [Result] Sohrabi C, Alsafi Z, O'Neill N, Khan M, Kerwan A, Al-Jabir A, Iosifidis C, Agha R. World Health Organization declares global emergency: A review of the 2019 novel coronavirus (COVID-19). Int J Surg. 2020 Apr;76:71-76. doi: 10.1016/j.ijsu.2020.02.034. Epub 2020 Feb 26. PMID 32112977
- [Result] Fu L, Wang B, Yuan T, Chen X, Ao Y, Fitzpatrick T, Li P, Zhou Y, Lin YF, Duan Q, Luo G, Fan S, Lu Y, Feng A, Zhan Y, Liang B, Cai W, Zhang L, Du X, Li L, Shu Y, Zou H. Clinical characteristics of coronavirus disease 2019 (COVID-19) in China: A systematic review and meta-analysis. J Infect. 2020 Jun;80(6):656-665. doi: 10.1016/j.jinf.2020.03.041. Epub 2020 Apr 10. PMID 32283155
- [Derived] Estebanez-Perez MJ, Martin-Valero R, Pastora-Estebanez P, Pastora-Bernal JM. Experiences of people with Long Covid with a digital physiotherapy intervention: A qualitative study. Health Expect. 2024 Apr;27(2):e13993. doi: 10.1111/hex.13993. PMID 38590093
- [Derived] Estebanez-Perez MJ, Pastora-Bernal JM, Vinolo-Gil MJ, Pastora-Estebanez P, Martin-Valero R. Digital physiotherapy is a satisfactory and effective method to improve the quality of life in Long COVID patients. Digit Health. 2024 Feb 26;10:20552076241234432. doi: 10.1177/20552076241234432. eCollection 2024 Jan-Dec. PMID 38414563
- [Derived] Estebanez-Perez MJ, Pastora-Bernal JM, Martin-Valero R. The Effectiveness of a Four-Week Digital Physiotherapy Intervention to Improve Functional Capacity and Adherence to Intervention in Patients with Long COVID-19. Int J Environ Res Public Health. 2022 Aug 3;19(15):9566. doi: 10.3390/ijerph19159566. PMID 35954922
- [Derived] Pastora-Bernal JM, Estebanez-Perez MJ, Molina-Torres G, Garcia-Lopez FJ, Sobrino-Sanchez R, Martin-Valero R. Telerehabilitation Intervention in Patients with COVID-19 after Hospital Discharge to Improve Functional Capacity and Quality of Life. Study Protocol for a Multicenter Randomized Clinical Trial. Int J Environ Res Public Health. 2021 Mar 12;18(6):2924. doi: 10.3390/ijerph18062924. PMID 33809277